CLINICAL TRIAL: NCT06056193
Title: SIRrolimus-coated Versus Plain Old Balloon Angioplasty (POBA) in Lower Extremity Autologous Venous Bypass Stenosis - The SIR-POBA Bypass Trial
Brief Title: The SIR-POBA Bypass Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited recruiting
Sponsor: Paracelsus Medical University (Other)
Collaborators: MedAlliance Swiss Medical Technology (Unknown)
Responsible Party: Principal Investigator, Manuela Pilz, Senior Physician, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1036/2023
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Arterial Occlusive Disease; Bypass Complication; Femoropopliteal Artery Occlusion; Femoropopliteal Stenosis; Critical Limb-Threatening Ischemia; Claudication, Intermittent
Keywords: Autologous Vein Bypass; Endovascular Revascularization
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Intermittent Claudication | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plain Balloon Angioplasty (Active Comparator): Plain Balloon Angioplasty will be used to treat lesions
  Interventions: Procedure: Balloon Angioplasty
- Sirolimus-coated Balloon Angioplasty (Active Comparator): Sirolimus-coated Balloon Angioplasty will be used to treat lesions after preparing vessel with plain balloon angioplasty
  Interventions: Procedure: Balloon Angioplasty

INTERVENTIONS:
Procedure: Balloon Angioplasty — Revascularisation procedures will be performed according to randomised list
  Other Names: Endovascular Revascularization

SUMMARY:
The goal of this clinical trial is to compare plain old balloon angioplasty with sirolimus-coated balloon angioplasty in patients with an infrainguinal venous bypass stenosis. The main question we aim to answer is, how patency is affected by each of the randomised treatment options.

DETAILED DESCRIPTION:
This clinical trial will be conducted at our Division of Vascular Surgery and Endovascular Surgery at the University Hospital of Salzburg. Patients will be randomized into one of the two treatment options (plain old ballon angioplasty versus sirolimus coated balloon angioplasty). The recruitment phase is calculated for two years with a planned follow-up of 2 years. Follow-up data will be collected to answer the endpoints and will include all available follow-ups to monitor the bypass up to 2 years after the procedure. Typically, follow-up visits will be conducted at 6 weeks, 3 months, 6 months, 12 months, and 24 months after the procedure.

ELIGIBILITY:
Inclusion Criteria

* Age at least 18 years
* Informed consent with signature
* Rutherford category 2 or 3 (in terms of lifestyle-limiting moderate or severe claudication symptomatology) or chronic critical ischemia (Rutherford 4-6)
* Venous bypass stenosis requiring intervention
* Confirmed inflow
* At least 1 crural outflow vessel

Exclusion Criteria:

* Pregnant or lactating women
* Active infection or sepsis
* Patients currently participating in another clinical trial
* Unconfirmed inflow
* Intolerance to sirolimus
* Coagulopathy
* Radiotherapy
* Patients on immunosuppressive therapy
* Non-dialysis renal insufficiency (eGFR < 45 ml/min/1.73m2)
* Use of potent CYP3A4 and/or P-gp inhibitors (such as ketoconazole, Voriconazole, itraconazole, erythromycin, telithromycin, or clarithromycin) or strong CYP3A4 and/or P-gp inducers (such as rifampin or rifabutin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Primary Lesion Target Patency of the venous bypass stenosis | 2 years
  The incidence of patency will be analysed after reopening the stenosis of the venous bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Pilz, MD PD FEBVS, Principal Investigator — Senior Physician; Klaus Linni, MD PD FEBVS, Study Director — Head of Division of Vascular and Endovascular Surgery; Stephanie Rassam, MD, Study Chair — Resident Physician
Locations (1):
- University Hospital of Salzburg, Paracelsus Medical University, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No